CLINICAL TRIAL: NCT04699136
Title: Use and Validation of the 6-minute Stepper Test in in Patients With Cardiac Pathologies Needing Rehabilitation and Reeducation (CVRR)
Brief Title: Cardiovascular Rehabilitation and Reeducation (CVRR) in Patients With Cardiac Pathologies and the 6-minute Stepper Test
Acronym: STEPPER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lille Catholic University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RC-P0087; 2019-A02483-54 (Other: IDRCB)
Record Dates: First submitted 2021-01-06; First posted 2021-01-07 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Cardiac Disease
Keywords: Cardiovascular rehabilitation; Stepper test; 6-minute
MeSH Terms: conditions — Heart Diseases | interventions — Exercise Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cardiovascular disease (Experimental)
  Interventions: Other: 6 minutes step test (ST6)

INTERVENTIONS:
Other: 6 minutes step test (ST6) — Performing a 6 minutes step test at different intervals and comparing with respect with the 6 minutes walk test and cardiac stress test

SUMMARY:
The objective is to study the validity of the 6-minute stepper test (ST6) in order to determine tolerance to effort in cardiovascular patients

DETAILED DESCRIPTION:
The 6-minute stepper test (ST6) is an test used and validated in patients with respiratory disorders (chronic obstructive pulmonary disease) in order to evaluate their tolerance to exercise. It is well tolerated and reproducible in these patients, with the advantage that it can be performed without spatial constraints.

However, this test is not yet used in cardiology. This study proposes to validate the ST6, to evaluate the exercise tolerance of patients suffering from cardiovascular pathologies.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old,
* Patient with a cardiac pathology (coronary bypass, valve replacement, heart transplant, coronary angioplasty),
* Registered in Cardiovascular Rehabilitation at the Mitterie Clinic,
* Number of rehabilitation sessions at least equal to 30,
* Ejection fraction ≥ 45%,
* Signed written consent of the patient,
* Affiliation to a social security scheme.

Exclusion Criteria:

* Cardiac decompensation,
* Severe functional limitation,
* Unstable acute coronary syndrome,
* Decompensated heart failure,
* Severe ventricular rhythm disorders,
* Presence of an intracardiac thrombus with high embolic risk,
* Presence of a medium to large pericardial effusion (effusion of more than 10mm circumferential or 14mm localized on ultrasound),
* Recent history (months prior to inclusion) of thrombophlebitis with or without pulmonary embolism,
* Severe and/or symptomatic left ventricular ejection obstruction,
* Any progressive inflammatory and/or infectious disease,
* Severe pulmonary arterial hypertension,
* Oxygen therapy,
* Musculoskeletal or balance problems that would limit the ability to do any of the following the fiscal year.
* Pregnant or breastfeeding women,
* Incapacity to consent (including persons under guardianship or curatorship)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-01-13 (Actual); Primary Completion 2022-04-28 (Actual); Study Completion 2022-04-28 (Actual)

PRIMARY OUTCOMES:
Internal validity of the 6 minutes step test (ST6) | Day 0
  The number of steps taken in 6 minutes with the ST6 will be measured twice on the first day of the cardiovascular rehabilitation and education. The second ST6 will be performed 30 minutes after the first. Internal validity will be studied by calculating the intra-class correlation coefficient (ICC) of the number of steps from the two ST6 carried out and its 95% confidence interval.
External validity of the ST6 with respect to the 6 minutes walk test (WT6) | Day 0
  The external validity with respect to the (6 minutes walk test) WT6 will be studied by calculating the Pearson correlation coefficient and its 95% confidence interval between the number of steps from the ST6 and the distance travelled in meters from the WT6.

SECONDARY OUTCOMES:
External validity of the ST6 with respect to the cardiac stress test | Day 0
  The external validity with respect to the cardiac stress test will be studied by calculating the Pearson correlation coefficient and its 95% confidence interval between the number of steps from the ST6 and the cardiac stress test.
External validity of the ST6 with respect to the Oxygen saturation at rest. | Day 0
  The external validity with respect to the Oxygen saturation at rest will be studied by calculating the Pearson correlation coefficient and its 95% confidence interval between the number of steps from the ST6 and the Oxygen saturation at rest.
External validity of the ST6 with respect to the heart rate at maximum effort | Day 0
  The external validity with respect to the heart rate at maximum effort will be studied by calculating the Pearson correlation coefficient and its 95% confidence interval between the number of steps from the ST6 and the heart rate.

CONTACTS AND LOCATIONS:
Overall Officials: Amandine SECQ, MD, Principal Investigator — Clinique de la Mitterie
Locations (1):
- Clinique de la Mitterie, Lille, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Racodon M, Fabre C, Vanhove P, Vale JD, Bolpaire R, Moutailler E, Malanda F, Secq A. Validity and Reproducibility of the Six-Minute Stepper Test in Cardiac Patients. J Cardiovasc Transl Res. 2025 Aug;18(4):993-1000. doi: 10.1007/s12265-025-10624-z. Epub 2025 May 8. PMID 40341471